CLINICAL TRIAL: NCT05195515
Title: The Impact of Late Effects After Treatment for Bladder Cancer on Quality of Life - What is the Cost of the Cure?
Brief Title: The Impact of Late Effects After Treatment for Bladder Cancer on Quality of Life
Acronym: CONQUER
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); National Research Center for Survivorship and Late Adverse Effects Following Pelvic Organ Cancer, Denmark (Unknown)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, DMSc, Aarhus University Hospital
Other Study IDs: CONQUER
Record Dates: First submitted 2022-01-07; First posted 2022-01-19 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Bladder Cancer
Keywords: Quality of Life; Bladder Cancer; Late effects
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder Cancer prognosis, treatment, and subsequent morbidity and mortality vary between the different stages, thus resulting in a different impact on patients' lives. There are some well known late effects of the treatments for bladder cancer, but the knowledge of their impact on patients Quality of Life is sparse. This study aims to determine the prevalence of late effects impact on Quality of Life and potential risk factors for impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are referred to a hospital in the Central Region Denmark, due to hematuria between 01/01/2022 and 01/01/2023
* Ability to understand written and oral Danish

Exclusion Criteria:

* Known Alzheimers disease
* Diagnosed other causes explaining the hematuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, referred due to hematuria
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life | 5 years from baseline inclusion
  Changes in Quality of Life measured using validated instruments

SECONDARY OUTCOMES:
Prevalence of late effects | 5 years from baseline inclusion
  Based on Patient Reported Outcomes and medical records

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Bjerggaard Jensen, Professor, Principal Investigator — Department of Urology, Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Department of Urology, Aarhus University Hospital, Aarhus N
  - Department of Urology, Regional Hospital Gødstrup, Gødstrup
  - Department of Urology, Regional Hospital Horsens, Horsens
  - Department of Urology, Regional Hospital Randers, Randers
  - Department of Urology, Regional Hospital Viborg, Viborg